CLINICAL TRIAL: NCT03327727
Title: A Phase 2 Study of VL-2397 Compared to Standard First-Line Treatment for Invasive Aspergillosis in Adults With Acute Myelogenous Leukemia, Acute Lymphocytic Leukemia, or Allogeneic Hematopoietic Cell Transplant Recipients
Brief Title: VL-2397 Compared to Standard First-Line Treatment for Invasive Aspergillosis (IA) in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Vical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VL2397-201; 2017-003435-11 (EudraCT Number)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Invasive Aspergillosis; Invasive Pulmonary Aspergillosis
Keywords: IA
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis | interventions — isavuconazole; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Sponsor, safety monitoring board, and data review committee are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VL-2397 (Experimental): Investigational agent VL-2397 600 mg IV infusion administered every day for 28 days (4 weeks) followed by 2 weeks of standard treatment
  Interventions: Drug: Investigational Agent: VL-2397; Drug: Standard treatment: Voriconazole, Isavuconazole, or Liposomal amphotericin B
- Standard (First-Line) Treatment (Active Comparator): Investigator selected standard treatments of voriconazole, isavuconazole, or liposomal amphotericin B administered every day for 42 days (6 weeks) per product package insert
  Interventions: Drug: Standard treatment: Voriconazole, Isavuconazole, or Liposomal amphotericin B

INTERVENTIONS:
Drug: Investigational Agent: VL-2397 — VL-2397
  Arms: VL-2397
Drug: Standard treatment: Voriconazole, Isavuconazole, or Liposomal amphotericin B — Voriconazole, Isavuconazole, or Liposomal amphotericin B

SUMMARY:
The purpose of the trial is to evaluate the safety and efficacy of a new antifungal with a novel mechanism of action in immunocompromised adults with invasive aspergillosis.

DETAILED DESCRIPTION:
To compare the safety and efficacy of VL-2397 to standard first-line treatment for invasive aspergillosis in immunocompromised adults with acute leukemia or recipients of an allogeneic hematopoietic cell transplant (allo-HCT).

ELIGIBILITY:
Inclusion Criteria:

* Acute Leukemia (AML or ALL) patient or allo-HCT recipient with a diagnosis of IA

Exclusion Criteria:

* Pregnant or breastfeeding
* IA involving sites other than lungs and sinuses
* Graft failure, acute or extensive chronic GvHD
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
All-cause mortality (ACM) | 4 weeks

SECONDARY OUTCOMES:
ACM | 6 weeks
Number of participants with adverse events | 6 weeks
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mammen P Mammen, MD, FIDSA, Study Director — Vical
Locations (28):
- United States (11):
  - University of Alabama at Birmingham Hospital, Division of Infectious Diseases, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Davis Health, Dept. of Internal Medicine, Div. of Infectious Diseases, Sacramento, California
  - Christiana Care Health Services, Department of Medicine, Newark, Delaware
  - Medical College of Georgia at Augusta University, Augusta, Georgia
  - DMC Harper University Hospital, Detroit, Michigan
  - University of Minnesota, Department of Medicine, Minneapolis, Minnesota
  - Washington University School of Medicine, Division of Infectious Disease, St Louis, Missouri
  - The University of Texas Health Science Center, Department of Internal Medicine, Houston, Texas
  - Fred Hutchinson Cancer Research Center (FHCRC), Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (5):
  - University Hospital Antwerp (UZA), Department of Hematology, Edegem, Antwerp
  - General Hospital Saint-Jan, Department of Hematology, Bruges
  - Jules Bordet Institute, Department of Infectious Disease, Brussels
  - University Hospitals Leuven, Campus Gasthuisberg, Department of Hematology, Leuven
  - UCL Mont-Godinne University Hospitals, Department of Hematology, Yvoir
- Canada (3):
  - Hamilton Health Sciences, Infectious Disease Research, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre (MUHC), Division of Infectios Diseases, Montreal, Quebec
- France (3):
  - Grenoble University Hospital Center, Department of Hematology, Grenoble
  - South Lyon Hospital Center, Pierre-Bénite
  - Hautepierre Hospital, Strasbourg
- Germany (2):
  - University Hospital Jena, Jena
  - Hospital Neuperlach - Municipal Hospital Munich GmbH, Clinic of Hematology and Oncology, Munich
- South Korea (4):
  - Chonnam National University, Hwasun
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No